CLINICAL TRIAL: NCT04236596
Title: Pudendal Nerve Mapping Towards Improved Neuromodulation for Urinary Retention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Timothy Bruns, Associate Professor of Biomedical Engineering, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00165005; OT2OD028191 (NIH)
Record Dates: First submitted 2020-01-13; First posted 2020-01-22 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Urinary Retention; Underactive Bladder
Keywords: pudendal nerve mapping
MeSH Terms: conditions — Urinary Retention; Urinary Bladder, Underactive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Study participants (Experimental): Study participants received an implanted neurostimulator at their pudendal nerve as part of normal clinical care. This was not an intervention study as clinical care was not modified based on study participation. Participants consented to undergo in the research study steps towards mapping of the pudendal nerve.
  Interventions: Device: Participants received a Neurostimulator, which was used to map the pudendal nerve

INTERVENTIONS:
Device: Participants received a Neurostimulator, which was used to map the pudendal nerve — Participants in study received neurostimulator at their pudendal nerve as part of their normal clinical care. This neurostimulator was used to map the nerve.

SUMMARY:
This study is to map the pudendal nerve. In this study the researchers will examine subjects who are already receiving an implanted stimulator at their pudendal nerve as part of their normal clinical care.

DETAILED DESCRIPTION:
The pudendal nerve goes to the urethra, anus, and other areas of the pelvic floor. Electrical stimulation of this nerve can help with bladder problems and pelvic pain. Researchers do not understand how the nerve anatomy is different between people. Successfully mapping the pudendal nerve may help improve the medical care for future patients with bladder problems, pelvic pain, bowel problems, and sexual problems.

ELIGIBILITY:
Inclusion Criteria:

* Clinically referred as having bladder problems that have not responded to conservative treatment. Normal clinical care includes referral to implant of Medtronic Interstim neurostimulator at the pudendal nerve. Fully eligible to receive an Interstim implant.
* Adult (18 or older), capable of providing own informed consent and communicating clearly with research team
* Capable of speaking, reading, and understanding English, as all study questionnaires are standardized assessments only available in English
* Capable of attending all experimental sessions (Visit 1: pre-stage-1 imaging, Visit 2: stage-1 surgery, Visit 3: CT after stage-2 surgery, Visit 3: cystometrogram test)

Exclusion

* Implanted materials that prohibit magnetic imaging
* Any medical problems that prevent an individual from laying flat in an MRI or CT scanner, are are claustrophobic.
* Areflexive or atonic bladder
* Pregnant or planning to become pregnant. If a woman of child-bearing potential wishes to participate in this study, they will be pre-screened with a test to detect pregnancy.
* Diagnosed neurogenic bladder, pudendal nerve damage, lower motor dysfunction, or other conditions that would affect the neural circuits involved in micturition.
* Unwilling to allow de-identified data to be stored for future use or shared with other researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Bruns, Ph.D., Principal Investigator — University of Michigan; Priyanka Gupta, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified IPD collected during the trial will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Will be available starting twelve months following publication of study findings.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Derived] Chen PJ, Lagunas AC, Soriano V, Gupta P, Bruns TM. Perineal and Rectal Nerve Recruitment Order Varies During Pudendal Neurostimulator Implant Surgery. Neurourol Urodyn. 2025 Apr;44(4):851-859. doi: 10.1002/nau.70010. Epub 2025 Feb 10. PMID 39927446

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Participants: Study participants are receiving an implanted neurostimulator at their pudendal nerve and consent to undergo study procedures.
Period: Overall Study
Arm/Group | Study Participants
Started | 22
Completed | 14
Not Completed | 8
Not completed — Withdrawal by Subject | 1
Not completed — Participants did not retain implant for entire trial | 3
Not completed — Participants did not receive implant at all | 4

BASELINE CHARACTERISTICS:
Groups:
- Study Participants: Study participants received an implanted neurostimulator at their pudendal nerve and consented to participate in study activities.
Arm/Group | Study Participants
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.37 (13.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Evoked Bladder Contractions of at Least 20 Centimeters of Water (cmH2O) During the Stage-4 Test
Description: The primary outcome measure in this study was an evoked bladder contraction of at least 20 centimeters of water (cmH2O) during the cystometrogram. These bladder contractions were evoked by applying nerve stimulation to the pudendal nerve through testing of the participant's implanted stimulator. Measure reflects number of participants who experienced an evoked bladder contraction of at least 20 centimeters of water during nerve stimulation.
Time Frame: Visit 4, approximately 10 weeks after consent
Population: Due to scheduling conflicts and participant attrition, only 10 participants completed this part of the study. All were women.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Undergoing Cystometrogram: This group includes participants who underwent the cystometrogram procedure.
Arm/Group | Participants Undergoing Cystometrogram
Number analyzed (Participants) | 10
Participants | 0

2. Secondary Outcome: Selectivity Index (SI) for Selective Stimulation of Pudendal Nerve Branches for Participant Stimulation
Description: Selectivity refers to the degree in which a nerve could be stimulated without stimulating other nerves. SI was calculated for each sensor recording from locations innervated by distal pudendal nerve branches during the visit-2 implant procedure. This includes pressure sensors in the urethra innervated by the perineal nerve and anal electromyography (EMG) innervated by the ischeal rectal nerve. The SI calculation used here is on a scale of 0 to 1, with 0 indicating no response at all from the nerve. The closer the number is to 1, the more selective the nerve stimulated.
Time Frame: Visit 2: Stage-1 (approximately 3 weeks after consent)
Population: Data was collected from 16 participants who received the implant.
Measure: Mean (Standard Deviation); unit: index
Groups:
- Participants Undergoing Stage-2 Implant Data Collection: These participants underwent the stage-2 data collection procedure and had functional sensor recordings during pudendal nerve stimulation, allowing for SI calculations.
Arm/Group | Participants Undergoing Stage-2 Implant Data Collection
Number analyzed (Participants) | 16
index
  Perineal nerve | 0.57 (0.29)
  Rectal nerve | 0.90 (0.22)

3. Secondary Outcome: Selectivity Index (SI) for Selective Stimulation of Pudendal Nerve Branches for Simulated Model Stimulation
Description: Selectivity is the degree to which part of a nerve could be stimulated without stimulating other nerve parts. For each participant who had successful MRI and CT images, a computational model was created to simulate electrical stimulation of axons distributed in two primary pudendal fascicles: perineal and rectal. The SI of stimulation does not indicate a positive or negative result in this outcome; rather, it shows the relative potential for activating just a single nerve fascicle. The negative/positive designation identifies the regional nerve activation, with -1 representing only perineal fascicle activation, +1 representing only rectal activation, and 0 indicating equal activation of both fascicles.
Time Frame: Approximately one year and four months after consent
Population: Computational models were created for 10 participants who received the implant. The model data was segregated into three groups: participants with selectivity indices positive (>0) for all four contacts (rectal only), negative (<0) for all four contacts (perineal only), and mixed (both >0 and <0). Each group has the same potential range for SI values: -1 to +1. Values in the Outcome Measure Data Table are calculations across all lead contacts and participants per group.
Measure: Mean (Standard Deviation); unit: index
Groups:
- Selectivity Index: Selectivity index calculation across all models (4 contacts per model)
Arm/Group | Selectivity Index
Number analyzed (Participants) | 10
index
  Rectal dominant: number analyzed (Participants) | 4
  Rectal dominant | 0.577 (0.193)
  Perineal dominant: number analyzed (Participants) | 3
  Perineal dominant | -0.533 (0.284)
  Mixed: number analyzed (Participants) | 3
  Mixed | 0.288 (0.666)

4. Secondary Outcome: Measurement of Effect of Pudendal Nerve Stimulation on Urethral Leak Point Pressure During the Stage-4 Test
Description: A secondary outcome measure was a goal to examine the effect of selective pudendal nerve stimulation on urethral leak point pressure during the cystometrogram.
Time Frame: Visit 4, approximately 10 weeks after consent
Population: Selective pudendal nerve stimulation was not performed during the cystometrogram sessions due to time limitations within experimental sessions, so there is no data available. "Selectivity" could not be accomplished as it was described in the protocol for this nerve bundle.
Arm/Group | Participants Undergoing Cystometrogram
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Approximately 2 years and 8 months
Arm/Group | Study Participants
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT04236596/Prot_000.pdf
  • Informed Consent Form (2023-09-24): https://cdn.clinicaltrials.gov/large-docs/96/NCT04236596/ICF_001.pdf